CLINICAL TRIAL: NCT06795126
Title: Augmented Reality for Managing Pediatric Anxiety and Pain During Disasters - A Randomized Pilot Feasibility Study
Brief Title: Little NIRVANA for Pediatric Pain and Anxiety
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: KU Leuven (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan Chang, Emergency Medicine Physician, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00004268; U1IMC43532 (Other Grant/Funding Number: Health Resources and Services Administration (HRSA))
Record Dates: First submitted 2025-01-22; First posted 2025-01-27 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-01

CONDITIONS: Acute Pain; Procedural Anxiety; Pediatric ALL; Emergency Medicine; IV Access
Keywords: AR; Pain; Anxiety; Augmented Reality; Distraction
MeSH Terms: conditions — Acute Pain; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive a topical anesthetic cream and will use Little NIRVANA AR digital solution during PIV line placement
  Interventions: Other: Little NIRVANA
- Control (No Intervention): Treatment as usual - participants will receive a topical anesthetic cream but will not use the Little NIRVANA (other distraction methods available in the ED are allowed)

INTERVENTIONS:
Other: Little NIRVANA — Augmented reality (AR) digital solution where children interact with the game using a magic wand
  Other Names: Augmented Reality
  Arms: Intervention Group

SUMMARY:
The aim of this study is to test the feasibility of using Little NIRVANA (augmented reality (AR)) for managing anxiety and pain for children 2-8 years old during hospital emergency peripheral intravenous (PIV) insertions. The investigators hypothesize that Little NIRVANA plus a numbing cream will reduce pain and anxiety for patients undergoing PIV placement in the emergency department (ED) when compared to the cream alone. It is anticipated that using the Little NIRVANA will not increase the ED length of stay, failed PIV placement attempts, or the need for additional intervention.

DETAILED DESCRIPTION:
This is a two-group randomized clinical trial of 65 dyads of subjects and their parent and 65 proceduralists. Children will be randomly assigned to either the Little NIRVANA intervention group or a standard of care control group. Legal guardians of children in both groups will answer questions about their child's prior history of needle procedures, current pain/anxiety, medications taken prior to ED arrival, and video game experience. Children assigned to the intervention will play the game during the PIV placement, while children in the control group will receive the standard of care. The proceduralist performing the PIV placement and the parent will answer questions after the PIV placement about their perception of the child's pain and anxiety and questions about the Little NIRVANA experience for those children who were in the intervention group. This study has one visit that is completed during their ED stay.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing PIV line placement (peripheral IV order placed while patient is in the ED);
* Patients 2-8 years of age (inclusive)

Exclusion Criteria:

* Non-English speaking (Little NIRVANA is currently only available in English and Dutch);
* those for whom utilizing AR is deemed not feasible by the attending ED physician (e.g., critical illness)

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proxy reported pain | Immediately following the PIV line placement
  0-10 Numerical Rating Scale (NRS) (proxy reported by parent and proceduralist), 0(minimum)-10(maximum), with higher score indicating worse pain.
Proxy reported anxiety | Immediately following the PIV line placement
  0-10 Numerical Rating Scale (NRS) (proxy reported by parent and proceduralist), 0(minimum )-10(maximum), with higher score indicating worse anxiety.

SECONDARY OUTCOMES:
Proxy reported AR experience | Immediately following the PIV line placement
  0-10 Numerical Rating Scale (NRS) (proxy-reported - intervention arm only), 0(minimum )-10(maximum), with higher score meaning better outcome. Asked for fun, engagement, and satisfaction with the AR.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No